CLINICAL TRIAL: NCT00762710
Title: Clinical Trial of the Adrenergic Alpha-1 Antagonist Prazosin for Alcohol Dependence
Brief Title: Study of the Medication Prazosin for Alcohol Dependence
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seattle Institute for Biomedical and Clinical Research (Other)
Collaborators: National Institute on Alcohol Abuse and Alcoholism (NIAAA) (NIH); VA Puget Sound Health Care System (U.S. Federal Agency); University of Washington (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1R01AA017184-01 (NIH); 5R01AA017184-05 (NIH)
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Alcoholism
Keywords: Alcohol; Abuse; Use; Disorder; Dependence; Symptoms; Alcoholic; Alcoholism; Prazosin; Drug; Medicine; Medication; Treatment; Study; Placebo; Medical; Management; Craving; Consumption; Binge; Drinking; Drink; Heavy
MeSH Terms: conditions — Alcoholism; Disease; Binge-Eating Disorder | interventions — Prazosin

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 - Prazosin Medication (Experimental): Following randomization, participants in this arm will receive a 2-week titration of Prazosin followed by 10 weeks of stable dosing of Prazosin. They will also attend study visits at least weekly for 12 weeks and will complete a final follow-up one month after discontinuation of the medication phase of the study at 16 weeks post-randomization.
  Interventions: Drug: Prazosin medication
- 2 - Placebo Medication (Placebo Comparator): Following randomization, participants in this arm will receive a 2-week titration of placebo followed by 10 weeks of stable dosing of placebo. They will also attend study visits at least weekly for 12 weeks and will complete a final follow-up one month after discontinuation of the medication phase of the study at 16 weeks post-randomization.
  Interventions: Drug: Placebo medication

INTERVENTIONS:
Drug: Prazosin medication — Form: Prazosin will be taken orally, in the form of pills.
  Dosing: 9 AM, 3 PM, 9 PM
  Days 1-2: 0 mg, 0 mg, 1 mg
  Days 3-4: 1 mg, 1 mg, 1 mg
  Days 5-7: 2 mg, 2 mg, 2 mg
  Day 8-10: 2 mg, 2 mg, 6 mg
  Day 11-14: 4 mg, 4 mg, 6 mg
  Day 15-84: 4 mg, 4 mg, 8 mg
  Other Names: Minipress
  Arms: 1 - Prazosin Medication
Drug: Placebo medication — Form: Placebo will be taken orally, in the form of pills.
  Dosing: 9 AM, 3 PM, 9 PM
  Days 1-2: 0 mg, 0 mg, 1 mg
  Days 3-4: 1 mg, 1 mg, 1 mg
  Days 5-7: 2 mg, 2 mg, 2 mg
  Day 8-10: 2 mg, 2 mg, 6 mg
  Day 11-14: 4 mg, 4 mg, 6 mg
  Day 15-84: 4 mg, 4 mg, 8 mg
  Other Names: No other intervention names
  Arms: 2 - Placebo Medication

SUMMARY:
The purpose of this study is to determine whether the drug prazosin is effective for the treatment of alcohol dependency.

DETAILED DESCRIPTION:
Alcohol dependence (AD) afflicts nearly 10% of the US population and causes marked medical morbidity and mortality, marked psychiatric morbidity, increased health care costs, and lost work hours (Saxon, Malte, Sloan, et al., 2006; McFall, Saxon, Thaneemit-Chen, et al., 2007). Alcohol dependence is a biologically, genetically based disease, yet the majority of clinically accepted treatments are behaviorally or psychosocially based (Anton, O'Malley, Ciraulo, et al., 2006; Todd, Armeli, Tennen, et al., 2005). Despite the initial success of these treatments, 40-70% of patients relapse within the first 12 months after treatment (McGinnis & Foege, 1993). Research is needed to develop more effective biological treatments.

Currently, only three pharmacological treatments are FDA approved for the treatment of alcohol dependence and all are sub-optimal. None of these medications directly target noradrenergic brain systems. Recent advances in understanding the neurobiology of substance dependence and relapse support the notion that adrenergic systems play a critical role in these processes.

In a 6-week, double-blind, placebo-controlled pilot study, we randomized 24 participants without PTSD entering treatment for AD to prazosin or identical appearing placebo (Simpson et al., 2009). The prazosin group reported no more adverse events than the placebo group, and controlling for drinks per week at baseline and week number, the prazosin group reported fewer drinks per week in the final 3 weeks of the study. These findings led us to conduct a larger trial to further evaluate prazosin for AD.

The current study is a 16-week, randomized, two group parallel-design, double-blind, placebo-controlled trial to evaluate the efficacy of prazosin for decreasing alcohol use and the subjective experience of alcohol craving in individuals without PTSD who are seeking treatment for AD. Following randomization, a 2-week titration period will be followed by 10 weeks of stable dosing of prazosin or placebo. Study participants will attend study visits at least weekly for 12 weeks and will complete a final follow-up one month after discontinuation of the medication phase of the study at 16 weeks post-randomization. All study participants will also participate in Medical Management (MM) treatment, a behavioral intervention that has demonstrated efficacy as a behavioral platform for treatment of AD (Anton, O'Malley, Ciraulo, et al., 2006). Study participants will not be involved in other professional counseling or substance abuse treatment during their study involvement, though 12-step meeting attendance is encouraged during MM. Daily monitoring of alcohol craving, alcohol use, other substance craving and substance use, medication compliance, and key psychiatric symptoms via toll-free telephone calls to an Interactive Voice Response (IVR) system will continue throughout the 16-week study. Outcome measures will address alcohol use and craving and include IVR reports of craving and use, the TLFB for alcohol use, Penn Alcohol Craving Scale (PACS), Patient Health Questionnaire-9 (depression), urine toxicology analysis (UDA), and Breathalyzer readings.

ELIGIBILITY:
Inclusion Criteria:

* Current primary DSM-IV diagnosis of alcohol dependence(AD)
* Heavy drinking in the last 30 days
* At least 18 years of age
* Good general medical health (see Exclusion Criteria below)
* Capacity to provide informed consent
* English fluency and literacy

Exclusion Criteria:

* Psychiatric/behavioral: current post-traumatic stress disorder(PTSD); psychiatric disorder requiring any medication other than anti-depressants; currently taking disulfiram, acamprosate, or naltrexone or planning to take any of these medications during the 12-week medication phase of the study; current dependence on any other psychoactive substance other than nicotine or cannabis; a current diagnosis of opioid abuse, use of any opioid- containing medications or benzodiazepines during the previous month, or UDA positive for opioids, benzodiazepines, or sedative hypnotics.
* Medical: significant acute or chronic medical illness; women who are pregnant, nursing infant(s), or of childbearing potential and not using a contraceptive method judged by the study physician or PA to be effective; signs or symptoms of alcohol withdrawal at the time of initial consent
* Legal involvement that could interfere with study treatment. Individuals court ordered for treatment will not be eligible to participate in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2008-01 (Actual); Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tracy L Simpson, Ph.D., Principal Investigator — VA Puget Sound Health Care System
Locations (1):
- VA Puget Sound Health Care System, Seattle, Washington, United States

REFERENCES:
- [Background] Saxon AJ, Malte CA, Sloan KL, Baer JS, Calsyn DA, Nichol P, Chapko MK, Kivlahan DR. Randomized trial of onsite versus referral primary medical care for veterans in addictions treatment. Med Care. 2006 Apr;44(4):334-42. doi: 10.1097/01.mlr.0000204052.95507.5c. PMID 16565634
- [Background] McFall M, Saxon AJ, Thaneemit-Chen S, Smith MW, Joseph AM, Carmody TP, Beckham JC, Malte CA, Vertrees JE, Boardman KD, Lavori PW. Integrating smoking cessation into mental health care for post-traumatic stress disorder. Clin Trials. 2007;4(2):178-89. doi: 10.1177/1740774507076923. PMID 17456521
- [Background] Anton RF, O'Malley SS, Ciraulo DA, Cisler RA, Couper D, Donovan DM, Gastfriend DR, Hosking JD, Johnson BA, LoCastro JS, Longabaugh R, Mason BJ, Mattson ME, Miller WR, Pettinati HM, Randall CL, Swift R, Weiss RD, Williams LD, Zweben A; COMBINE Study Research Group. Combined pharmacotherapies and behavioral interventions for alcohol dependence: the COMBINE study: a randomized controlled trial. JAMA. 2006 May 3;295(17):2003-17. doi: 10.1001/jama.295.17.2003. PMID 16670409
- [Background] Todd M, Armeli S, Tennen H, Carney MA, Ball SA, Kranzler HR, Affleck G. Drinking to cope: a comparison of questionnaire and electronic diary reports. J Stud Alcohol. 2005 Jan;66(1):121-9. doi: 10.15288/jsa.2005.66.121. PMID 15830912
- [Background] McGinnis JM, Foege WH. Actual causes of death in the United States. JAMA. 1993 Nov 10;270(18):2207-12. PMID 8411605
- [Derived] Simpson TL, Saxon AJ, Stappenbeck C, Malte CA, Lyons R, Tell D, Millard SP, Raskind M. Double-Blind Randomized Clinical Trial of Prazosin for Alcohol Use Disorder. Am J Psychiatry. 2018 Dec 1;175(12):1216-1224. doi: 10.1176/appi.ajp.2018.17080913. Epub 2018 Aug 29. PMID 30153753

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in January 2008 and ended June 2014. Six hundred and one people responding to flyers and newspaper advertisements and contacted the study, 151 provided informed consent, and 19 women and 73 men (N = 92) were randomized. Both civilian and veteran participants were seen in an outpatient VA clinic.
Pre-assignment Details: Of the 151 consented into the study, 59 did not go onto be randomized because of the following:
  Declined after screen (N=11) (includes missing baseline/first medication appointment) Ineligible at screen (N=48)
  * PTSD (N=11)
  * Acute illness (N=7)
  * Drug dependence (N=4)
  * Drinking inclusion not met (N=20)
  * Other (N=6)
Groups:
- Prazosin: Prazosin medication
  Prazosin medication: Form: Prazosin will be taken orally, in the form of pills.
  Dosing: 9 AM, 3 PM, 9 PM
  Days 1-2: 0 mg, 0 mg, 1 mg
  Days 3-4: 1 mg, 1 mg, 1 mg
  Days 5-7: 2 mg, 2 mg, 2 mg
  Day 8-10: 2 mg, 2 mg, 6 mg
  Day 11-14: 4 mg, 4 mg, 6 mg
  Day 15-84: 4 mg, 4 mg, 8 mg
- Placebo: Placebo medication
  Placebo medication: Form: Placebo will be taken orally, in the form of pills.
  Dosing: 9 AM, 3 PM, 9 PM
  Days 1-2: 0 mg, 0 mg, 1 mg
  Days 3-4: 1 mg, 1 mg, 1 mg
  Days 5-7: 2 mg, 2 mg, 2 mg
  Day 8-10: 2 mg, 2 mg, 6 mg
  Day 11-14: 4 mg, 4 mg, 6 mg
  Day 15-84: 4 mg, 4 mg, 8 mg
Period: Overall Study
Arm/Group | Prazosin | Placebo
Started | 48 | 44
Completed | 27 | 29
Not Completed | 21 | 15

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Prazosin | Placebo | Total
Number analyzed (Participants) | 48 | 44 | 92
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 48 | 44 | 92
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (9.8) | 49.1 (9.5) | 48.1 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 8 | 19
  Male | 37 | 36 | 73
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 48 | 44 | 92

OUTCOME MEASURES:

1. Primary Outcome: Alcohol Consumption
Description: At the baseline and final medication visits, the Form 90 (19) was used to assess alcohol and drug use for the preceding 90-day period
Time Frame: 12 weeks
Population: Providing baseline and last week of medication information for all participants that completed the titration period (40 in each group).
Measure: Mean (Standard Deviation); unit: percentage of days heavy drinking
Arm/Group | Prazosin | Placebo
Number analyzed (Participants) | 40 | 40
percentage of days heavy drinking
  Baseline % Days Heavy Drinking | 71.8 (29.1) | 66.5 (26.0)
  Final medication week % Days Heavy Drinking | 11.4 (22.8) | 22.6 (34.1)

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events after they started taking medications and about one month after they discontinued the medications. Because a few participants withdrew from the study after the baseline, where medications were dispensed, adverse events were monitored from one week to 16 weeks, depending on the length of participants' participation in the study.
Description: Participants were queried at every study visit with regard to potential adverse events and underwent clinical safety checks (e.g., sitting and stand blood pressures) at each visit.
Arm/Group | Prazosin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/48 | 1/44
Serious Adverse Events (participants affected / at risk) | 3/48 | 2/44
Other Adverse Events (participants affected / at risk) | 28/48 | 15/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Prazosin (N=48) | Placebo (N=44)
Death (Psychiatric disorders) | 0 (0) | 1 (1) — Placebo participant committed suicide.
Medical hospitalization (Infections and infestations) | 1 (1) | 0 (0) — prazosin participant admitted to hospital for infected wisdom tooth
medical hospitalization (Gastrointestinal disorders) | 0 (0) | 1 (1) — placebo participant hospitalized for acute pancreatitis
inpatient alcohol detoxification (Psychiatric disorders) | 2 (2) | 0 (0) — two prazosin participants were hospitalized for acute alcohol withdrawal
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Prazosin (N=48) | Placebo (N=44)
Drowsiness (General disorders) | 28 | 15

LIMITATIONS AND CAVEATS:
Lack of knowledge of optimal dosing for prazosin and medication adherence (medication adherence was suboptimal).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Informed Consent Form (2013-09-09): https://cdn.clinicaltrials.gov/large-docs/10/NCT00762710/ICF_000.pdf